CLINICAL TRIAL: NCT05913401
Title: Aerobic Exercise to Augment the Plasticity Effect of rTMS in Patients With Treatment-resistant Depression
Brief Title: Exercise to Augment TMS in Those With Treatment Resistant Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2304-001; P20GM130452 (NIH)
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Treatment Resistant Depression
Keywords: Aerobic Exercise; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise (Experimental): Exercise sessions will be 20 minutes of moderate-intensity aerobic exercise on a treadmill. A treadmill is located on D1A within the space shared by the Butler Hospital TMS Clinic and the COBRE-support Neuromodulation Research Facility. A research staff member will monitor their heart rate and blood pressure to ensure safety and that activity is occurring at a moderate intensity (i.e., 64-76% of age predicted maximal heart rate). Participants will be asked to rate their affect and rating of perceived exertion (RPE) during exercise sessions. Sessions will include a 5-min warm-up and a 5-min cool-down to ensure safe exercise procedures. Participants will be asked to answer questions about affect before, during, and after exercise. These sessions will be supervised (i.e., they provide onsite coverage) by an exercise physiologist or medical staff member (e.g., nurse or physician) to ensure safety.
  Interventions: Behavioral: Aerobic Exercise
- Video Condition (Other): In this condition, participants will be asked to sit and watch various documentaries or educational videos on topics NOT related to physical activity. These will last approximately 20 minutes and will occur before each TMS session.
  Interventions: Behavioral: Video Watching

INTERVENTIONS:
Behavioral: Aerobic Exercise — 20 minutes of supervised aerobic exercise on a treadmill prior to each TMS session
  Arms: Aerobic Exercise
Behavioral: Video Watching — 20 minutes of watching documentaries or educational videos prior to each TMS session
  Arms: Video Condition

SUMMARY:
Given the growing evidence that aerobic increases cortical excitability and promotes neuroplasticity, the scientific premise for its potential priming effect on the brain is strong. Combining AE with rTMS may produce a neural environment optimized for a robust physiological effect of rTMS, thereby leading to improved depression outcomes. With positive findings, this study would provide preliminary support for an innovative, safe and feasible approach for improving outcomes for this significant public health problem.

DETAILED DESCRIPTION:
Depression is highly prevalent and a significant public health concern, resulting in tremendous economic and societal burden. With first-line treatments leaving the majority of patients with unremitted and impairing symptomatology, additional therapies to address treatment-resistant depression (TRD) are critical. One such approach that has received significant empirical attention is repetitive transcranial magnetic stimulation (rTMS). While effective in reducing depression, rTMS's efficacy is not without limits, with remission rates being less than 40%. Therefore, research focused on improving the efficacy of rTMS is timely and critical for decreasing the overall public health burden of TRD. A putative mechanism of the effect of rTMS on depression is through changes in electrophysiological properties of neurons leading to increases in long-term potentiation (LTP) necessary for neuroplasticity. In theory, it may be possible to improve rTMS outcomes by augmenting it with another non-pharmacological treatment known to influence neuroplasticity. One innovative possibility could be aerobic exercise (AE), as it has shown to result in increased neuroplasticity in both animal and human studies and is known to reduce depression. There are a number of neural effects of AE that could serve to prime the brain for rTMS including increased prefrontal oxygenation and increased brain-derived neurotropic factor (BDNF, involved in inducing LTP). Conceivably, bouts of AE just prior to rTMS sessions may create a neural environment that is broadly primed for the more focally delivered TMS, potentially increasing its effectiveness. To date, there have been no studies that have combined AE with rTMS. Therefore, the purpose of the proposed study is to conduct the first test of AE priming among treatment-resistant depressed individuals seeking rTMS treatment. We expect that AE will improve the efficacy of rTMS through changes in exercise-induced neuroplasticity via measurements of motor-evoked potential (MEP). Exercise studies have shown single bouts of aerobic activity can result in increased MEP amplitudes and chronic AE (i.e., multi-sessions) decreases resting motor thresholds (RMT; the lowest intensity of TMS that evokes a MEP), thereby increasing overall cortical excitability. For the proposed pilot study, we will recruit N=30 patients with treatment-resistant depression who are seeking rTMS treatment at Butler Hospital's TMS Clinic. Participants will be randomized to engage in one of two different activities just prior to their scheduled daily TMS treatments: 1) 20 minutes of supervised moderate-intensity AE on an on-site treadmill (n=15) OR 2) 20-minutes of watching an educational video (n=15) while sitting. To examine indicators of neuroplasticity, a TMS cortical excitability protocol (assessing plasticity through measuring MEPs generated by single and paired magnetic pulses) will be conducted at baseline (prior to initiating the course of rTMS) and then again after 30 rTMS treatment sessions. At these same timepoints, depression severity will be measured using the Inventory of Depressive Symptomatology-Self Report scale (IDS-SR). The feasibility and acceptability of the combined AE+TMS approach will also be examined to inform the design of a future larger trial.

ELIGIBILITY:
Inclusion Criteria:

* adult outpatients (age 18 and above) who are already approved to receive standard TMS therapy through the Butler Hospital TMS clinic.
* able to safely engage in moderate-intensity aerobic exercise (determined by a study physician)

Exclusion Criteria:

* Currently pregnant or plans to become pregnant in the next 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Intervention Acceptability | Baseline
  Percentage of participants approached for the study who agree to participate
Feasibility of Intervention | 6-weeks
  Percentage of sessions attended (out of a possible 30 sessions)

SECONDARY OUTCOMES:
Resting state motor thresholds | 6-weeks
  A measure of corticolspinal excitation
short-interval intracortical inhibition (SICI) | 6-weeks
  A measure of GABAa channel activity
short-interval intracortical facilitation (SICF) | 6-weeks
  A reflection of glutamatergic tone uninhibited by GABA interneurons

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
Data will be made available to other researchers upon request.